CLINICAL TRIAL: NCT02186600
Title: Randomized Control Trial of Bone Loading Exercises Versus Risedronate on Bone Health in Post-Menopausal Women
Brief Title: Heartland Osteoporosis Prevention Study
Acronym: HOPS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Nebraska (Other)
Collaborators: Creighton University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0378-14-FB
Record Dates: First submitted 2014-07-07; First posted 2014-07-10 (Estimated); Results first posted 2023-06-27 (Actual); Last update posted 2023-10-05 (Actual); Status verified 2023-09

CONDITIONS: Osteopenia
Keywords: Low bone mass; Post-menopausal women; Bone mineral density; Bone structure; Bone turnover; Bone-loading exercises; calcium and vitamin D; risedronate
MeSH Terms: conditions — Bone Diseases, Metabolic | interventions — Calcium Carbonate; Drugs, Generic; Cholecalciferol; Risedronic Acid

STUDY DESIGN:
Intervention Model Description: Randomized to 3 treatment groups: Calcium + vitamin D only; risedronate and calcium + vitamin D; bone building exercises and calcium + vitamin D
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Control (Active Comparator): Women randomized to the control group will receive calcium and vitamin D intake for 12 months. Calcium intake will be determined by analyzing 3 day dietary intake of calcium at baseline and then prescribing calcium carbonate supplements to ensure women have ~1200 mg of calcium daily. Vitamin D intake will be determined using baseline measures of Serum 25 (OH) D. Subjects who have serum D levels of 30 ng/ml or greater will be prescribed 1,000 IU vitamin D3 daily; subjects with levels of 20-29 ng/ml will be prescribed 2,000 IU Vitamin D3; and subjects with levels of 10-19 ng/ml will be prescribed 3,000 IU Vitamin D3.
  Interventions: Drug: Calcium Carbonate; Drug: Vitamin D3
- Risedronate (Experimental): Subjects in the risedronate group will take 35 mg of the bisphosphonate "risedronate" weekly for 12 months plus CaD. They will be asked to follow the protocol for administration of risedronate including taking the medication upon arising in the morning with an 8 ounce glass of water, remaining upright for at least 30 minutes, and having no oral intake except water for at least 30 minutes.
  Interventions: Drug: Calcium Carbonate; Drug: Vitamin D3; Drug: Risedronate
- Exercise (Experimental): Subjects in the exercise group will participate in bone-loading exercises three times weekly in addition to taking CaD for 12 months. Women will exercise at community Young Men's Christian Association's fitness centers (YMCA) and exercises will be monitored by on-site Exercise Trainers. Exercises will consist of high-impact weight-bearing exercises (jogging with weighted vests) and resistance exercises for upper and lower extremities. Progressive increases in weight loads will be prescribed to provide maximal strength gains.
  Interventions: Drug: Calcium Carbonate; Drug: Vitamin D3; Behavioral: Bone-loading exercises

INTERVENTIONS:
Drug: Calcium Carbonate — Used as daily supplement to ensure subject obtains 1200 mg of calcium per day (diet + supplement)
  Other Names: generic
Drug: Vitamin D3 — Subjects will receive Vitamin D3 supplements to ensure serum level of Vitamin D is at least 30 ng/ml.
  Other Names: generic
Drug: Risedronate — Risedronate 35 mg orally will be ingested weekly by subjects in Risedronate group.
  Other Names: Actonel
  Arms: Risedronate
Behavioral: Bone-loading exercises — Subjects will participate in bone loading exercises (weight-bearing and resistance) three times weekly at community YMCAs.
  Arms: Exercise

SUMMARY:
The purpose of this study is to identify the best way to prevent bone loss in the first years after menopause. The HOPS study will compare bone loss at 12 months in women: 1) who take calcium and vitamin D only; 2) who take calcium and vitamin D plus the medication "risedronate"; or 3) who take calcium and vitamin D plus participate in bone-loading exercises. Our central hypothesis is that improvements in bone health will be greater in women randomized to bone-loading exercises with calcium and vitamin D compared to women who take calcium and vitamin D only or women who take calcium and vitamin D plus risedronate.

DETAILED DESCRIPTION:
This randomized controlled trial (RCT) will compare changes after 12 months in bone structure, bone mineral density (BMD), and bone turnover in women with low bone mass who are within 5 years of menopause. Women will be randomized to one control and 2 treatment groups (n =103 per group): 1) calcium + vitamin D (CaD) alone (Control); 2) Bisphosphonate (BP) plus optimal CaD (Risedronate); and 3) a bone loading exercise program plus optimal CaD (Exercise). Our central hypothesis is that improvements in bone health will be greater in subjects randomized to the exercise group compared to subjects in either the control or risedronate groups. Specific Aims: Aims 1, 2, and 3 are to compare control, risedronate, and exercise group subjects on changes in bone structure at the tibia and hip (measured by pQCT and Hip Structural Analysis) (Aim 1) ; on changes in BMD at the total hip, femoral neck, and spine (Aim 2); and on changes in serum markers of bone formation and resorption (Aim 3). In addition, Aim 4 will explore relationships between adherence to exercise (% sessions attended) or adherence to risedronate (% pills taken) and changes in bone structure.

ELIGIBILITY:
Inclusion Criteria:

* Women who are in their first 5 years of menopause
* Have a T score between -1 and -2.49 at the femoral neck, total hip, or L1-L4 spine
* Be 19 years of age or older
* Have their health care provider's permission to enroll in the study.

Exclusion Criteria:

* Have osteoporosis
* Have a 10 yr probability of hip fracture >3% or major fracture >20% based on results of the fracture risk assessment (FRAX) tool
* Currently take bisphosphonates, estrogen replacement therapy, glucocorticosteroids, or other drugs affecting bone
* Currently participate in a resistance training or high impact weight bearing exercise program three or more times weekly
* Weigh >300 lbs
* Have abnormal results for the following laboratory tests: serum 25(OH)D; serum creatinine; serum calcium; parathyroid hormone (PTH); thyroid stimulating hormone (TSH).
* Have Paget's disease, heart disease, uncontrolled hypertension, renal disease, or other concomitant conditions that prohibit participation in exercises, risedronate therapy, or use of CaD supplements.

Min Age: 19 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 276 (Actual)
Dates: Start 2015-02-01 (Actual); Primary Completion 2019-06-01 (Actual); Study Completion 2019-06-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nancy L Waltman, PhD, APRN-NP, Principal Investigator — University of Nebraska; Laura Bilek, PT, PhD, Principal Investigator — University of Nebraska
Locations (1):
- University of Nebraska Medical Center, Omaha, Nebraska, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bocalini DS, Serra AJ, dos Santos L, Murad N, Levy RF. Strength training preserves the bone mineral density of postmenopausal women without hormone replacement therapy. J Aging Health. 2009 Jun;21(3):519-27. doi: 10.1177/0898264309332839. Epub 2009 Feb 27. PMID 19252142
- [Background] Uusi-Rasi K, Kannus P, Cheng S, Sievanen H, Pasanen M, Heinonen A, Nenonen A, Halleen J, Fuerst T, Genant H, Vuori I. Effect of alendronate and exercise on bone and physical performance of postmenopausal women: a randomized controlled trial. Bone. 2003 Jul;33(1):132-43. doi: 10.1016/s8756-3282(03)00082-6. PMID 12919708
- [Background] Bergstrom I, Landgren B, Brinck J, Freyschuss B. Physical training preserves bone mineral density in postmenopausal women with forearm fractures and low bone mineral density. Osteoporos Int. 2008 Feb;19(2):177-83. doi: 10.1007/s00198-007-0445-6. Epub 2007 Sep 1. PMID 17768587
- [Background] Dane C, Dane B, Cetin A, Erginbas M. Effect of risedronate on biochemical marker of bone resorption in postmenopausal women with osteoporosis or osteopenia. Gynecol Endocrinol. 2008 Apr;24(4):207-13. doi: 10.1080/09513590801895617. PMID 18382907
- [Background] Cussler EC, Going SB, Houtkooper LB, Stanford VA, Blew RM, Flint-Wagner HG, Metcalfe LL, Choi JE, Lohman TG. Exercise frequency and calcium intake predict 4-year bone changes in postmenopausal women. Osteoporos Int. 2005 Dec;16(12):2129-41. doi: 10.1007/s00198-005-2014-1. Epub 2005 Nov 10. PMID 16283062
- [Background] Elders PJ, Netelenbos JC, Lips P, van Ginkel FC, Khoe E, Leeuwenkamp OR, Hackeng WH, van der Stelt PF. Calcium supplementation reduces vertebral bone loss in perimenopausal women: a controlled trial in 248 women between 46 and 55 years of age. J Clin Endocrinol Metab. 1991 Sep;73(3):533-40. doi: 10.1210/jcem-73-3-533. PMID 1874931
- [Background] Valimaki MJ, Farrerons-Minguella J, Halse J, Kroger H, Maroni M, Mulder H, Munoz-Torres M, Saaf M, Snorre Ofjord E. Effects of risedronate 5 mg/d on bone mineral density and bone turnover markers in late-postmenopausal women with osteopenia: a multinational, 24-month, randomized, double-blind, placebo-controlled, parallel-group, phase III trial. Clin Ther. 2007 Sep;29(9):1937-49. doi: 10.1016/j.clinthera.2007.09.017. PMID 18035193
- [Background] Vainionpaa A, Korpelainen R, Sievanen H, Vihriala E, Leppaluoto J, Jamsa T. Effect of impact exercise and its intensity on bone geometry at weight-bearing tibia and femur. Bone. 2007 Mar;40(3):604-11. doi: 10.1016/j.bone.2006.10.005. Epub 2006 Nov 30. PMID 17140871
- [Background] Waltman NL, Twiss JJ, Ott CD, Gross GJ, Lindsey AM, Moore TE, Berg K, Kupzyk K. The effect of weight training on bone mineral density and bone turnover in postmenopausal breast cancer survivors with bone loss: a 24-month randomized controlled trial. Osteoporos Int. 2010 Aug;21(8):1361-9. doi: 10.1007/s00198-009-1083-y. Epub 2009 Oct 3. PMID 19802506
- [Background] Fogelman I, Ribot C, Smith R, Ethgen D, Sod E, Reginster JY. Risedronate reverses bone loss in postmenopausal women with low bone mass: results from a multinational, double-blind, placebo-controlled trial. BMD-MN Study Group. J Clin Endocrinol Metab. 2000 May;85(5):1895-900. doi: 10.1210/jcem.85.5.6603. PMID 10843171
- [Background] Going S, Lohman T, Houtkooper L, Metcalfe L, Flint-Wagner H, Blew R, Stanford V, Cussler E, Martin J, Teixeira P, Harris M, Milliken L, Figueroa-Galvez A, Weber J. Effects of exercise on bone mineral density in calcium-replete postmenopausal women with and without hormone replacement therapy. Osteoporos Int. 2003 Aug;14(8):637-43. doi: 10.1007/s00198-003-1436-x. Epub 2003 Jul 3. PMID 12844212
- [Background] Kemmler W, Engelke K, Lauber D, Weineck J, Hensen J, Kalender WA. Exercise effects on fitness and bone mineral density in early postmenopausal women: 1-year EFOPS results. Med Sci Sports Exerc. 2002 Dec;34(12):2115-23. doi: 10.1097/00005768-200212000-00038. PMID 12471325
- [Background] Vainionpaa A, Korpelainen R, Vaananen HK, Haapalahti J, Jamsa T, Leppaluoto J. Effect of impact exercise on bone metabolism. Osteoporos Int. 2009 Oct;20(10):1725-33. doi: 10.1007/s00198-009-0881-6. Epub 2009 Mar 5. PMID 19262975
- [Background] Klentrou P, Slack J, Roy B, Ladouceur M. Effects of exercise training with weighted vests on bone turnover and isokinetic strength in postmenopausal women. J Aging Phys Act. 2007 Jul;15(3):287-99. doi: 10.1123/japa.15.3.287. PMID 17724395
- [Background] Prentice RL, Pettinger MB, Jackson RD, Wactawski-Wende J, Lacroix AZ, Anderson GL, Chlebowski RT, Manson JE, Van Horn L, Vitolins MZ, Datta M, LeBlanc ES, Cauley JA, Rossouw JE. Health risks and benefits from calcium and vitamin D supplementation: Women's Health Initiative clinical trial and cohort study. Osteoporos Int. 2013 Feb;24(2):567-80. doi: 10.1007/s00198-012-2224-2. Epub 2012 Dec 4. PMID 23208074
- [Background] Somford MP, Geurts GF, den Teuling JW, Thomassen BJ, Draijer WF. Long-Term Alendronate Use Not without Consequences? Int J Rheumatol. 2009;2009:253432. doi: 10.1155/2009/253432. Epub 2010 Jan 27. PMID 20148064
- [Background] Whyte MP. Atypical femoral fractures, bisphosphonates, and adult hypophosphatasia. J Bone Miner Res. 2009 Jun;24(6):1132-4. doi: 10.1359/jbmr.081253. PMID 19113923
- [Background] Caulfield MP, Reitz RE. Biochemical markers of bone turnover and their utility in osteoporosis. MLO Med Lab Obs. 2004 Apr;36(4):34-7. No abstract available. PMID 15119056
- [Background] Bischoff-Ferrari HA, Giovannucci E, Willett WC, Dietrich T, Dawson-Hughes B. Estimation of optimal serum concentrations of 25-hydroxyvitamin D for multiple health outcomes. Am J Clin Nutr. 2006 Jul;84(1):18-28. doi: 10.1093/ajcn/84.1.18. PMID 16825677
- [Background] Bischoff-Ferrari HA, Willett WC, Wong JB, Giovannucci E, Dietrich T, Dawson-Hughes B. Fracture prevention with vitamin D supplementation: a meta-analysis of randomized controlled trials. JAMA. 2005 May 11;293(18):2257-64. doi: 10.1001/jama.293.18.2257. PMID 15886381
- [Background] Ott SM. Long-term safety of bisphosphonates. J Clin Endocrinol Metab. 2005 Mar;90(3):1897-9. doi: 10.1210/jc.2005-0057. No abstract available. PMID 15758064
- [Background] Schneider JP. Should bisphosphonates be continued indefinitely? An unusual fracture in a healthy woman on long-term alendronate. Geriatrics. 2006 Jan;61(1):31-3. No abstract available. PMID 16405362
- [Background] Hamdy RC, Petak SM, Lenchik L; International Society for Clinical Densitometry Position Development Panel and Scientific Advisory Committee. Which central dual X-ray absorptiometry skeletal sites and regions of interest should be used to determine the diagnosis of osteoporosis? J Clin Densitom. 2002;5 Suppl:S11-8. doi: 10.1385/jcd:5:3s:s11. PMID 12464707
- [Background] van der Linden JC, Weinans H. Effects of microarchitecture on bone strength. Curr Osteoporos Rep. 2007 Jun;5(2):56-61. doi: 10.1007/s11914-007-0003-3. PMID 17521506
- [Background] Akhter MP, Lappe JM, Davies KM, Recker RR. Transmenopausal changes in the trabecular bone structure. Bone. 2007 Jul;41(1):111-6. doi: 10.1016/j.bone.2007.03.019. Epub 2007 Apr 10. PMID 17499038
- [Background] Beck TJ. Extending DXA beyond bone mineral density: understanding hip structure analysis. Curr Osteoporos Rep. 2007 Jun;5(2):49-55. doi: 10.1007/s11914-007-0002-4. PMID 17521505
- [Background] Twiss JJ, Waltman NL, Berg K, Ott CD, Gross GJ, Lindsey AM. An exercise intervention for breast cancer survivors with bone loss. J Nurs Scholarsh. 2009 Mar;41(1):20-7. doi: 10.1111/j.1547-5069.2009.01247.x. PMID 19335674
- [Background] Management of osteoporosis in postmenopausal women: 2010 position statement of The North American Menopause Society. Menopause. 2010 Jan-Feb;17(1):25-54; quiz 55-6. doi: 10.1097/gme.0b013e3181c617e6. PMID 20061894
- [Background] Lappe JM, Davies KM, Travers-Gustafson D, Heaney RP. Vitamin D status in a rural postmenopausal female population. J Am Coll Nutr. 2006 Oct;25(5):395-402. doi: 10.1080/07315724.2006.10719551. PMID 17031008
- [Background] Borah B, Dufresne TE, Chmielewski PA, Johnson TD, Chines A, Manhart MD. Risedronate preserves bone architecture in postmenopausal women with osteoporosis as measured by three-dimensional microcomputed tomography. Bone. 2004 Apr;34(4):736-46. doi: 10.1016/j.bone.2003.12.013. PMID 15050906
- [Background] Kanis JA, Hans D, Cooper C, Baim S, Bilezikian JP, Binkley N, Cauley JA, Compston JE, Dawson-Hughes B, El-Hajj Fuleihan G, Johansson H, Leslie WD, Lewiecki EM, Luckey M, Oden A, Papapoulos SE, Poiana C, Rizzoli R, Wahl DA, McCloskey EV; Task Force of the FRAX Initiative. Interpretation and use of FRAX in clinical practice. Osteoporos Int. 2011 Sep;22(9):2395-411. doi: 10.1007/s00198-011-1713-z. Epub 2011 Jul 21. PMID 21779818
- [Background] Garber CE, Blissmer B, Deschenes MR, Franklin BA, Lamonte MJ, Lee IM, Nieman DC, Swain DP; American College of Sports Medicine. American College of Sports Medicine position stand. Quantity and quality of exercise for developing and maintaining cardiorespiratory, musculoskeletal, and neuromotor fitness in apparently healthy adults: guidance for prescribing exercise. Med Sci Sports Exerc. 2011 Jul;43(7):1334-59. doi: 10.1249/MSS.0b013e318213fefb. PMID 21694556
- [Background] Maddalozzo GF, Widrick JJ, Cardinal BJ, Winters-Stone KM, Hoffman MA, Snow CM. The effects of hormone replacement therapy and resistance training on spine bone mineral density in early postmenopausal women. Bone. 2007 May;40(5):1244-51. doi: 10.1016/j.bone.2006.12.059. Epub 2006 Dec 29. PMID 17291843
- [Background] Ashe MC, Gorman E, Khan KM, Brasher PM, Cooper DM, McKay HA, Liu-Ambrose T. Does frequency of resistance training affect tibial cortical bone density in older women? A randomized controlled trial. Osteoporos Int. 2013 Feb;24(2):623-32. doi: 10.1007/s00198-012-2000-3. Epub 2012 May 12. PMID 22581292
- [Result] Waltman N, Kupzyk KA, Flores LE, Mack LR, Lappe JM, Bilek LD. Bone-loading exercises versus risedronate for the prevention of osteoporosis in postmenopausal women with low bone mass: a randomized controlled trial. Osteoporos Int. 2022 Feb;33(2):475-486. doi: 10.1007/s00198-021-06083-2. Epub 2021 Sep 14. PMID 34519832
- [Derived] Bilek LD, Waltman NL, Lappe JM, Kupzyk KA, Mack LR, Cullen DM, Berg K, Langel M, Meisinger M, Portelli-Trinidad A, Lang M. Protocol for a randomized controlled trial to compare bone-loading exercises with risedronate for preventing bone loss in osteopenic postmenopausal women. BMC Womens Health. 2016 Aug 30;16(1):59. doi: 10.1186/s12905-016-0339-x. PMID 27576310

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Control | Risedronate | Exercise
Started | 93 | 91 | 92
Completed | 77 | 78 | 72
Not Completed | 16 | 13 | 20

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | Risedronate | Exercise | Total
Number analyzed (Participants) | 93 | 91 | 92 | 276
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.34 (3.30) | 54.53 (3.07) | 54.47 (3.11) | 54.4 (3.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 93 | 91 | 92 | 276
  Male | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 11 | 12 | 31
  Not Hispanic or Latino | 85 | 80 | 80 | 245
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1 | 2
  Asian | 1 | 5 | 2 | 8
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 2 | 2 | 1 | 5
  White | 89 | 84 | 88 | 261
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Family History of Low Bone Mass or Osteoporosis [Count of Participants; unit: Participants] — Number of participants with a positive family history of osteoporosis.
  Participants | 57 | 52 | 53 | 162

OUTCOME MEASURES:

1. Primary Outcome: Change in Bone Strength Index of the Distal Tibia Based on Randomization to Control, Risedronate, or Exercise Group.
Description: Change in Bone Strength Index (BSI) of the distal tibia based on randomization to Control, Risedronate, or Exercise group.
  BSI (mg2/mm4) at the 4% tibial site will be measured using peripheral quantitative computed tomography (pQCT).
Time Frame: Baseline, 6, and 12 months
Population: Intent-to-treat
Measure: Mean (Standard Deviation); unit: mg^2/mm^4
Arm/Group | Control | Risedronate | Exercise
Number analyzed (Participants) | 93 | 91 | 92
mg^2/mm^4
  Baseline: number analyzed (Participants) | 85 | 85 | 87
  Baseline | 2098.7 (334.7) | 1993.3 (292.3) | 2001 (332.1)
  6 Months: number analyzed (Participants) | 78 | 77 | 73
  6 Months | 2105.89 (322.822) | 1997.32 (307.103) | 1987.42 (300.136)
  12 Months: number analyzed (Participants) | 72 | 70 | 67
  12 Months | 2107.2 (326.4) | 2014.2 (306.7) | 2009.2 (280.4)
Statistical Analysis 1: Comparison: Control vs Risedronate vs Exercise; Test type: Other — Hierarchical linear modeling for intent-to-treat analysis to analyze time X group interactions, adjusted for baseline total body lean mass and height; p = 0.7, hierarchical linear modeling; controlled for total lean mass and height

2. Secondary Outcome: Change in Bone Mineral Density (BMD) at the Spine (L1-L4) Based on Randomization to Control, Risedronate, or Exercise Group.
Description: Bone mineral density is the gold standard for diagnosis of low bone mass and osteoporosis and will be measured at the spine using Dual Energy X-ray Absorptiometry (DXA).
Time Frame: Baseline,6, and 12 months
Population: Intent to treat analysis
Measure: Mean (Standard Deviation); unit: g/cm^2
Arm/Group | Control | Risedronate | Exercise
Number analyzed (Participants) | 93 | 91 | 92
g/cm^2
  Baseline | 0.889 (0.076) | 0.892 (0.06) | 0.886 (0.064)
  6 Months: number analyzed (Participants) | 86 | 82 | 82
  6 Months | .887 (.0755) | .907 (.0666) | .878 (.0619)
  12 Months | 0.885 (0.070) | 0.911 (0.070) | 0.885 (0.065)
Statistical Analysis 1: Comparison: Control vs Risedronate vs Exercise; Test type: Other — hierarchical linear modeling; p = 0.01, hierarchical linear modeling

3. Secondary Outcome: Change in Serum Measures of Bone Resorption (Serum NTx) Based on Randomization to Control, Risedronate, or Exercise Group.
Description: Bone turnover is the process of removing old bone (resorption by osteoclasts) and replacing it with new bone (formation by osteoblasts). Menopause results in a brief period (~5 years) of accelerated turnover with resorption far exceeding formation. In this study, resorption will be measured by Serum NTx.
Time Frame: Baseline, 6, 12 months
Population: Intention to treat for persons who had valid data at baseline
Measure: Mean (Standard Deviation); unit: nanoMolar Bone Collagen Equivalents/L
Arm/Group | Control | Risedronate | Exercise
Number analyzed (Participants) | 80 | 78 | 77
nanoMolar Bone Collagen Equivalents/L
  Baseline | 13.99 (4.22) | 14.31 (4.44) | 15.03 (5.45)
  6 Months | 12.16 (3.84) | 10.30 (3.93) | 13.36 (5.83)
  12 Months | 12.36 (3.48) | 11.42 (4.71) | 13.92 (5.84)
Statistical Analysis 1: Comparison: Control vs Risedronate vs Exercise; Test type: Other — Hierarchical linear modeling; p < 0.007, hierarchical linear modeling

ADVERSE EVENTS:
Time Frame: 12 months for each participant
Description: At each study visit, participants were asked if they had any new health conditions or events. We had questionnaires that evaluated tolerance to the treatments which allowed us to communicate with those who experienced symptoms as a result of the intervention.
Arm/Group | Control | Risedronate | Exercise
All-Cause Mortality (participants affected / at risk) | 0/93 | 0/91 | 0/92
Serious Adverse Events (participants affected / at risk) | 0/93 | 0/91 | 0/92
Other Adverse Events (participants affected / at risk) | 9/93 | 30/91 | 4/92
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control (N=93) | Risedronate (N=91) | Exercise (N=92)
Constipation (Gastrointestinal disorders) | 9 (9) | 13 (13) | 2 (2)
Gi disturbances (Gastrointestinal disorders) | 0 (0) | 4 (4) | 0 (0)
muscle or joint pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 11 (11) | 2 (2)
Chest Pain or Dizziness (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2015-06-17): https://cdn.clinicaltrials.gov/large-docs/00/NCT02186600/Prot_SAP_000.pdf
  • Informed Consent Form (2020-01-27): https://cdn.clinicaltrials.gov/large-docs/00/NCT02186600/ICF_001.pdf